CLINICAL TRIAL: NCT03298555
Title: A Smartphone Application (HealthyMoms) to Promote Healthy Weight Gain, Diet and Physical Activity During Pregnancy: a Randomized Controlled Trial
Brief Title: The HealthyMoms Trial to Promote Healthy Gestational Weight Gain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Marie Löf, docent, Senior researcher, associate professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2016-01147
Record Dates: First submitted 2017-09-25; First posted 2017-10-02 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Gestational Mothers; Weight Gain
MeSH Terms: conditions — Weight Gain

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile phone based intervention (Experimental): This group will receive the smartphone app HealthyMoms between gestational week 14 and 37. The app will contain information and support to achieve a healthy weight gain and lifestyle during pregnancy. This group will also receive standard care.
  Interventions: Behavioral: Mobile phone based intervention
- Control (No Intervention): This group will only receive standard care.

INTERVENTIONS:
Behavioral: Mobile phone based intervention — Participants in the intervention group will receive a 6-month mobile phone based program via a mobile phone application specifically designed for this study. The program will include information, advice and strategies to promote healthy gestational weight gain.
  Arms: Mobile phone based intervention

SUMMARY:
Excessive gestational weight gain is a major public health problem. Traditional face-to-face intervention programs has been shown to be succesful in order to promote healthier weight gains, however, they are time-consuming and expensive. The objectives of this study are to assess whether a 6-month smartphone application can promote healthy gestational weight gain, dietary habits and physical activity in pregnant women.

DETAILED DESCRIPTION:
Excessive gestational weight gain (GWG) increases risks for pregnancy complications, postpartum weight retention and offspring obesity. Traditional intervention programs are time and cost intensive. Mobile technology (mHealth) has been successful for weight loss and behavior changes; however, their use in pregnancy need to be further examined. This study aims to evaluate the impact of a smartphone application (app) intervention on GWG, diet, physical activity and glucose homeostasis.

HealthyMoms is a randomized controlled trial recruiting women at the first maternity clinic visit (week 6-10) in the Linköping area, Sweden. Women will be randomized to the control or intervention group (n=150 per group). All women will receive standard care. The intervention group will also receive the HealthyMoms smartphone app promoting healthy eating, activity and GWG during 6 months. Pregnancy outcomes are GWG (primary), food intake (web-based questionnaire), fat mass (BodPod), glucose homeostasis, activity (accelerometer) in week 37. Maternal and infant body fatness will be assessed one week post partum.

ELIGIBILITY:
Inclusion Criteria:

* a single pregnancy
* aged 18 years or above
* be able to speak and read Swedish sufficiently well.

Exclusion Criteria:

* previous diagnosed eating disorder
* pre-pregnancy diabetes or medical conditions or pharmacological treatments prior to pregnancy that may affect body weight

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 305 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-11-04 (Actual)

PRIMARY OUTCOMES:
Gestational weight gain | At the end of the intervention which is 23 weeks after baseline
  Body weight in gestational week 37 minus body weight in gestational week 14

SECONDARY OUTCOMES:
Body fatness using air-displacement plethysmography | At the end of the intervention which is 23 weeks after baseline
  Body fatness in gestational week 37 minus body fatness in gestational week 14
Physical activity using accelerometry | At the end of the intervention which is 23 weeks after baseline
  Moderate-to-vigorous physical activity (MVPA) in gestational week 37 minus MVPA in gestational week 14. MVPA will be assessed using wrist-worn accelerometry (Actigraph wGT3x) during 7 days at both time points.
Diet quality using a web-based questionnaire | At the end of the intervention which is 23 weeks after baseline
  Diet quality in gestational week 37 minus diet quality in gestational week 14. Diet quality will be assessed using a web-based questionnaire (a combination of a food-frequency questionnaire and two 24 hour recalls)
Glycemia | At the end of the intervention which is 23 weeks after baseline
  Plasma glucose levels in gestational week 37 minus plasma glucose levels in gestational week 14
Maternal body fatness post partum | One week post partum
  Maternal body fatness 1 week post partum
Infant body fatness | One week of age
  Infant body fatness at 1 week of age

CONTACTS AND LOCATIONS:
Overall Officials: Marie Löf, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sandborg J, Migueles JH, Soderstrom E, Blomberg M, Henriksson P, Lof M. Physical Activity, Body Composition, and Cardiometabolic Health during Pregnancy: A Compositional Data Approach. Med Sci Sports Exerc. 2022 Dec 1;54(12):2054-2063. doi: 10.1249/MSS.0000000000002996. Epub 2022 Sep 3. PMID 36069838
- [Derived] Henriksson P, Migueles JH, Soderstrom E, Sandborg J, Maddison R, Lof M. User engagement in relation to effectiveness of a digital lifestyle intervention (the HealthyMoms app) in pregnancy. Sci Rep. 2022 Aug 13;12(1):13793. doi: 10.1038/s41598-022-17554-9. PMID 35963935
- [Derived] Sandborg J, Soderstrom E, Henriksson P, Bendtsen M, Henstrom M, Leppanen MH, Maddison R, Migueles JH, Blomberg M, Lof M. Effectiveness of a Smartphone App to Promote Healthy Weight Gain, Diet, and Physical Activity During Pregnancy (HealthyMoms): Randomized Controlled Trial. JMIR Mhealth Uhealth. 2021 Mar 11;9(3):e26091. doi: 10.2196/26091. PMID 33704075
- [Derived] Sandborg J, Henriksson P, Larsen E, Lindqvist AK, Rutberg S, Soderstrom E, Maddison R, Lof M. Participants' Engagement and Satisfaction With a Smartphone App Intended to Support Healthy Weight Gain, Diet, and Physical Activity During Pregnancy: Qualitative Study Within the HealthyMoms Trial. JMIR Mhealth Uhealth. 2021 Mar 5;9(3):e26159. doi: 10.2196/26159. PMID 33666554